CLINICAL TRIAL: NCT03091413
Title: Correlation Between Pi Max and Diaphragm Maximum Inspiratory Excursion Detected With Ultrasound During Weaning
Status: Withdrawn | Type: Observational
Why Stopped: not recruitment
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Candelaria de Haro, MD, Corporacion Parc Tauli
Other Study IDs: ECO-MIP
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Weaning; Diaphragm Ultrasound; Maximum Inspiratory Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- case group: diaphragm ultrasounds during weaning and Pimax measures
  Interventions: Diagnostic Test: diaphragm ultrasound

INTERVENTIONS:
Diagnostic Test: diaphragm ultrasound — For each patient intubated and ventilated in our ICU we will performed diaphragm ultrasound during the weaning process.
  We will performed the measurement of diaphragmatic maximum excursion during a maximal inspiration using an abdominal standard preset with M-mode, with the so called anatomical M-mode.
  We will put the probe in the right subcostal window to use the hepatic window to assess the movement of the diaphragm. We will performed the measure of the diaphragm excursion with patient in semi-recumbent position and through a transhepatic transverse oblique scan while the patient is on mechanical ventilation and undergo a Pimax maneuver, that consists in a temporary occlusion of the airway with an expiratory pause.
  We will performed the measure three times, and we will take into account the best one made by the patient.

SUMMARY:
This study evaluates the correlation between maximum inspiratory pressure (Pi max) and the diaphragm maximum inspiratory excursion measured with ultrasound during the weaning from invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Invasive Mechanical Ventilation > 24 hours.
* Readiness for weaning (following clinician decision made according to recent guidelines).

Exclusion Criteria:

* Impossibility to perform an echography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ICU patients of Hospital de Sabadell who meet criteria for weaning will be included in the study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pimax and diaphragm inspiratory excursion | 4 months
  To assess the correlation between maximum inspiratory pressure (Pi max) and the diaphragm maximum inspiratory excursion measured with ultrasound.

SECONDARY OUTCOMES:
Predicting value of diaphragm excursion | 4 months
  To assess the predicting value of the diaphragm maximum inspiratory excursion measured with ultrasound for the weaning success.
Combination index prediction for weaning | 4 months
  To assess if the diaphragm maximum inspiratory excursion measured with ultrasound alone or in combination with other index (RSBI, Δtdi%) can predict the weaning success.

CONTACTS AND LOCATIONS:
Locations (1):
- Candelaria De Haro, Sabadell, Barcelona, Spain